CLINICAL TRIAL: NCT01522326
Title: Acute Mountain Sickness Treatment: A Double-blind Comparison of Metoclopramide vs. Ibuprofen
Brief Title: Comparison of Metoclopramide and Ibuprofen for the Treatment of Acute Mountain Sickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, N. Stuart Harris MD MFA, Director, MGH Wilderness Medicine Fellowship; Chief, Division of Wilderness Medicine, Department of Emergency Medicine, Massachusetts General Hospital; Assistant Professor of Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010P002837
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Acute Mountain Sickness; High Altitude Headache
Keywords: Acute Mountain Sickness; High Altitude Headache; Lake Louise AMS Score; Visual Analog Scale; Ibuprofen; Metoclopramide; Nepal
MeSH Terms: conditions — Altitude Sickness | interventions — Ibuprofen; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoclopramide (Experimental): 150 subjects with acute mountain sickness will be randomly assigned to take metoclopramide.
  Interventions: Drug: Metoclopramide
- Ibuprofen (Active Comparator): 150 subjects with acute mountain sickness will be randomly assigned to take ibuprofen.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 400mg tablet. Take one dose by mouth.
  Other Names: Advil; Motrin
  Arms: Ibuprofen
Drug: Metoclopramide — Metoclopramide 10mg tablet. Take one tablet by mouth.
  Other Names: Reglan
  Arms: Metoclopramide

SUMMARY:
The objective of this study is to determine the efficacy of metoclopramide in relieving the symptoms of Acute Mountain Sickness (AMS).

It is our hypothesis that the combined antiemetic and analgesic effects of metoclopramide (which has been study-proven to be effective in relieving symptoms of migraine headache) will prove to be more efficacious in relieving symptoms of acute mountain sickness than the standard, previously-studied analgesic medication, ibuprofen.

DETAILED DESCRIPTION:
Acute Mountain Sickness (AMS) is a well described disease process that occurs as a result of rapid exposure to high altitude. High altitude headache (HAH) is defined as the presence of headache in the setting of a recent increase in altitude. When HAH is associated with nausea, vomiting, fatigue, weakness, dizziness, lightheadedness or poor sleeping, AMS is diagnosed. While benign, AMS is very common, afflicting up to 80 % of travelers who ascend rapidly to 14,000 ft, and can be debilitating. AMS is thought to occur secondary to hypoxia-induced cerebral vasodilation. The antiemetic metoclopramide has been well studied and is commonly administered for treatment of migraine headaches in emergency departments across the U.S. The symptoms of migraine headaches are often similar to those of AMS. The mechanism of metoclopramide"s beneficial effect in this indication appear to be a result of its antagonism of central and peripheral dopamine receptors,most notably by blocking stimulation of the medullary chemoreceptor trigger zone. No studies have yet evaluated the potential benefits of metoclopramide for the relief of AMS. In contrast, ibuprofen has been well studied and found to be an effective treatment for the relief of symptoms of high altitude headache and AMS.

The study will be a convenience sample of trekkers traveling through the Annapurna Circuit in Nepal during the 3 month time period of March-May, 2012. Subjects will be recruited from visitors to Manang, Nepal staying in local hostels, those visiting the Himalayan Rescue Association clinic in Manang, and those responding to locally posted signage regarding study enrollment.

Eligible patients will be consented and enrolled in the study. Patients will be randomized to receive either Ibuprofen 400mg or Metoclopramide 10mg by mouth. Investigators will be blinded as to which arm of the study the patient is enrolled. Participants will be assessed by Lake Louise Score and Visual Analog Scale for headache and nausea severity immediately prior to ingestion of study medication, and then serially at 30, 60, and 120 minutes following medication ingestion. Standard statistical analysis of the Lake Louise AMS scores and visual analog scales will be used to determine which medication is more effective in treating acute mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* Presence at Manang recruitment center (at approximately 11,500 ft) during the dates March through May, 2012.
* Recent increase in altitude of > 1000 ft vertical in last 24 hours
* Presence of headache and at least one other symptom required for diagnosis of acute mountain sickness (including nausea, vomiting, fatigue, weakness, dizziness, lightheadedness or poor sleeping.)

Exclusion Criteria:

* Age less than 19 years old
* Known allergy or contraindication to either ibuprofen or metoclopramide
* Evidence of severe high altitude illness (e.g. High altitude pulmonary edema (HAPE) as evidenced by dyspnea at rest -- or of High Altitude Cerebral Edema (HACE) as evidenced by altered mental status or ataxia)
* Known or suspected pregnancy
* Use of other analgesic or antiemetic within 8 hours of study enrollment
* History of migraines or other chronic headache disorders
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-03-01; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Headache and Nausea Visual Analog Scales | 120 minutes
  Subjects will complete 100mm visual analog scales of both headache and nausea at time zero, 30, 60, and 120 minutes after taking the study medication. Visual analog scales are a valid assessment of symptom severity for acute mountain sickness.

SECONDARY OUTCOMES:
Lake Louise Acute Mountain Sickness Score | 120 minutes
  Subjects will take the Lake Louise Acute Mountains Sickness score before taking the medication and 120 minutes after taking the medication. The Lake Louise Acute Mountain Sickness Score is a standard measure of the severity of acute mountain sickness and is commonly used in studies involving acute mountain sickness.

CONTACTS AND LOCATIONS:
Overall Officials: Norman S Harris, MD, MFA, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Manang Clinic of the Himalayan Rescue Association, Manang, District of Manang, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roach RC, Bartsch P, Hackett PH, Oelz O. The Lake Louise acute mountain sickness scoring system. Hypoxia and Molecular Medicine, J.R. Sutton, C. S. Huston, and G. Coates eds. Burlinton, VT, USA: Queen City Printers; 1993.
- [Background] Gilbert DL. The first documented report of mountain sickness: the China or Headache Mountain story. Respir Physiol. 1983 Jun;52(3):315-26. doi: 10.1016/0034-5687(83)90088-9. PMID 6351209
- [Background] Gilbert DL. The first documented description of mountain sickness: the Andean or Pariacaca story. Respir Physiol. 1983 Jun;52(3):327-47. doi: 10.1016/0034-5687(83)90089-0. PMID 6351210
- [Background] Hultgren HN. High Altitude Pulmonary Edema. High Altitude Medicine. Stanford, CA: Hultgren Publications; 1997.
- [Background] Montgomery AB, Mills J, Luce JM. Incidence of acute mountain sickness at intermediate altitude. JAMA. 1989 Feb 3;261(5):732-4. PMID 2911169
- [Background] Maggiorini M, Buhler B, Walter M, Oelz O. Prevalence of acute mountain sickness in the Swiss Alps. BMJ. 1990 Oct 13;301(6756):853-5. doi: 10.1136/bmj.301.6756.853. PMID 2282425
- [Background] Schneider M, Bernasch D, Weymann J, Holle R, Bartsch P. Acute mountain sickness: influence of susceptibility, preexposure, and ascent rate. Med Sci Sports Exerc. 2002 Dec;34(12):1886-91. doi: 10.1097/00005768-200212000-00005. PMID 12471292
- [Background] Hackett PH, Roach RC. High-altitude illness. N Engl J Med. 2001 Jul 12;345(2):107-14. doi: 10.1056/NEJM200107123450206. No abstract available. PMID 11450659
- [Background] Ellsworth AJ, Meyer EF, Larson EB. Acetazolamide or dexamethasone use versus placebo to prevent acute mountain sickness on Mount Rainier. West J Med. 1991 Mar;154(3):289-93. PMID 2028586
- [Background] Zell SC, Goodman PH. Acetazolamide and dexamethasone in the prevention of acute mountain sickness. West J Med. 1988 May;148(5):541-5. PMID 3051673
- [Background] Hackett PH, Rennie D, Levine HD. The incidence, importance, and prophylaxis of acute mountain sickness. Lancet. 1976 Nov 27;2(7996):1149-55. doi: 10.1016/s0140-6736(76)91677-9. PMID 62991
- [Background] Broome JR, Stoneham MD, Beeley JM, Milledge JS, Hughes AS. High altitude headache: treatment with ibuprofen. Aviat Space Environ Med. 1994 Jan;65(1):19-20. PMID 8117220
- [Background] Gertsch JH, Lipman GS, Holck PS, Merritt A, Mulcahy A, Fisher RS, Basnyat B, Allison E, Hanzelka K, Hazan A, Meyers Z, Odegaard J, Pook B, Thompson M, Slomovic B, Wahlberg H, Wilshaw V, Weiss EA, Zafren K. Prospective, double-blind, randomized, placebo-controlled comparison of acetazolamide versus ibuprofen for prophylaxis against high altitude headache: the Headache Evaluation at Altitude Trial (HEAT). Wilderness Environ Med. 2010 Sep;21(3):236-43. doi: 10.1016/j.wem.2010.06.009. Epub 2010 Jun 16. PMID 20832701
- [Background] Harris NS, Wenzel RP, Thomas SH. High altitude headache: efficacy of acetaminophen vs. ibuprofen in a randomized, controlled trial. J Emerg Med. 2003 May;24(4):383-7. doi: 10.1016/s0736-4679(03)00034-9. PMID 12745039
- [Background] Kirthi V, Derry S, Moore RA, McQuay HJ. Aspirin with or without an antiemetic for acute migraine headaches in adults. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD008041. doi: 10.1002/14651858.CD008041.pub2. PMID 20393963
- [Background] Griffith JD, Mycyk MB, Kyriacou DN. Metoclopramide versus hydromorphone for the emergency department treatment of migraine headache. J Pain. 2008 Jan;9(1):88-94. doi: 10.1016/j.jpain.2007.09.001. Epub 2007 Nov 5. PMID 17981511
- [Background] Friedman BW, Corbo J, Lipton RB, Bijur PE, Esses D, Solorzano C, Gallagher EJ. A trial of metoclopramide vs sumatriptan for the emergency department treatment of migraines. Neurology. 2005 Feb 8;64(3):463-8. doi: 10.1212/01.WNL.0000150904.28131.DD. PMID 15699376
- [Background] Colman I, Brown MD, Innes GD, Grafstein E, Roberts TE, Rowe BH. Parenteral metoclopramide for acute migraine: meta-analysis of randomised controlled trials. BMJ. 2004 Dec 11;329(7479):1369-73. doi: 10.1136/bmj.38281.595718.7C. Epub 2004 Nov 18. PMID 15550401
- [Background] The Lake Louise Consensus on the Definition and Quantification of Altitude Illness. In: Sutton J, Coates G, Houston C, eds. Hypoxia and Molecular Medicine. Burlington, VT: Queen City Printers; 1993.
- [Background] Kayser B, Aliverti A, Pellegrino R, Dellaca R, Quaranta M, Pompilio P, Miserocchi G, Cogo A. Comparison of a visual analogue scale and Lake Louise symptom scores for acute mountain sickness. High Alt Med Biol. 2010 Spring;11(1):69-72. doi: 10.1089/ham.2009.1046. PMID 20367491